CLINICAL TRIAL: NCT03333356
Title: Adjuvant Radiotherapy in Patients With Pathological High-risk Bladder Cancer: A Randomized Multicentre Phase II Study
Brief Title: Adjuvant Radiotherapy in Patients With Pathological High-risk Bladder Cancer (GETUG-AFU 30)
Acronym: Bladder-ART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UC-0160/1617; 2016-A01535-46 (Registry Identifier: ANSM)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Patients With High-risk MIBC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): adjuvant pelvic radiotherapy consisting of 28 x 1.8 Gy fractions (total dose of 50.4 Gy), 5 days per week, 1 fraction / day (duration of RT is 38 days).
  Interventions: Radiation: pelvic radiotherapy
- Standard Arm (No Intervention): Surveillance

INTERVENTIONS:
Radiation: pelvic radiotherapy — adjuvant pelvic radiotherapy consisting of 28 x 1.8 Gy fractions (total dose of 50.4 Gy), 5 days per week, 1 fraction / day (duration of RT is 38 days).
  Arms: Experimental Arm

SUMMARY:
This is a randomized multicentre study in patients with high-risk MIBC to investigate adjuvant radiotherapy after radical cystectomy and pelvic lymph node dissection.

The objective of the study is to provide evidence that adjuvant radiotherapy improves loco-regional control with potential benefits in survival. The study will also evaluate the quality of life of patients and the tolerance of the treatment.

DETAILED DESCRIPTION:
INDICATION:

Patients with pathological high-risk muscle invasive bladder cancer treated by radical cystectomy and pelvic lymph nodes dissection

METHODOLOGY:

Multicenter randomised phase II study in high-risk bladder cancer patients treated by radical cystectomy with pelvic lymph nodes dissection assessing :

* Experimental Arm: adjuvant pelvic radiotherapy consisting of 28 x 1.8 Gy fractions (total dose of 50.4 Gy), 5 days per week, 1 fraction /day (duration of RT is 38 days).
* Standard Arm: surveillance. Eligible patients will be randomised, in a 3:1 ratio, to receive either: adjuvant pelvic radiotherapy (Experimental Arm), or surveillance (Standard Arm).

PRIMARY OBJECTIVE:

The primary objective of the trial is to assess the efficacy of adjuvant radiotherapy in patients with high-risk bladder cancer after radical cystectomy and pelvic lymph nodes dissection. Efficacy will be assessed in terms of pelvic recurrence-free survival (PRFS) at 3 years.

SECONDARY OBJECTIVES:

For each treatment arm (adjuvant pelvic radiotherapy [Experimental Arm], or surveillance [Standard Arm]), these objectives will be evaluated independently.

* To evaluate 5-year pelvic recurrence-free survival (PRFS)
* To evaluate disease-free survival (DFS) at 3 and 5 years.
* To evaluate overall survival (OS) at 3 and 5 years.
* To evaluate metastasis-free survival (MFS) at 3 and 5 years.
* To evaluate disease-specific survival (DSS) at 3 and 5 years.
* To evaluate the tolerance and safety of each treatment strategy.
* To evaluate patients' quality of life.

Ancillary studies Objectives:

* Investigation of individual predisposition to develop radiotherapy induced late digestive toxicity using the radiation-induced lymphocyte apoptosis (RILA) assay
* The analyse of genomic and transcriptome correlation between different clusters and oncological outcomes
* Dosimetric banking to evaluate the correlation of Dose-Volume Histogram with:
* Gastrointestinal toxicity grade ≥2;
* Pelvic recurrence (radiotherapy volumes, mapping of recurrences).

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the patients must fulfil all of the following inclusion criteria:

1. Patients with histologically-confirmed muscle-invasive bladder cancer, either with pure urothelial carcinomas, or dominant urothelial carcinomas (>50%) combined with other histological variants including: micropapillary, epidermoid, or adenocarcinomas, are eligible. Patients with small cell variants, pure adenocarcinomas, or pure epidermoid carcinomas are not eligible.
2. Patients with radical cystectomy and pelvic lymph nodes dissection with no microscopic residual disease (R0 and R1).

   Note that only R1 patients without urinary diversion as orthotropic neo-bladder replacement are eligible for the study, to limit cystectomy bed radiation induced toxicities.
3. Patients with tumours of TNM staging: pN0-2, M0 by imagery, and pT3a, pT3b, pT4a, and pT4b, as well as, pTX-pN1-2, pTX-NX-R1 are eligible.
4. Patients having received neo-adjuvant or adjuvant chemotherapy treatment are eligible. Randomization is allowed only if AE due to chemotherapy are ≤grade 2 at randomization.
5. Patients ≥18 years old.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Absolute neutrophil count (ANC) ≥1500 cells/mm³.
8. Platelets ≥100000 cells/mm³.
9. Haemoglobin ≥8 g/dL (Note: following a blood transfusion or another intervention if required).
10. Adequate hepatic function: aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤2.5 x upper limit of normal (ULN); or ≤3.5 x ULN in the case of concurrent disease with known etiology and for which a corrective treatment is possible.
11. Adequate renal function: clearance >30 mL/min (MDRD).
12. Patients having provided written informed consent prior to any study-related procedures.
13. Patients affiliated to the social security scheme.
14. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.

Exclusion Criteria:

Patient must not be enrolled if he/she fulfils any of the following non-inclusion criteria:

1. Patients with R1 resection and with orthotropic neo-bladder reconstruction as urinary diversion are not eligible.
2. Patients with clinical or radiological evidence of metastases or N3 staged bladder cancer are not eligible.
3. Prior invasive solid tumours or haematological malignancies unless disease free for a minimum of 3 years prior to randomisation except:

   * skin basal cell carcinoma,
   * in situ epithelioma of the cervix,
   * or prostate cancer: incidentally discovered during cystoprostatectomy and pelvic lymph node dissection and with a good prognosis (T stage <pT3b and/or Gleason <8 and pN- and/or post-operative prostate-specific antigen (PSA) <0.1 nanogram/mL),
4. Prior pelvic radiotherapy.
5. Patients with active inflammatory bowel disease.
6. Patients who required surgical treatment for bowel obstruction before bladder cancer diagnosis or after cystectomy.
7. Prior chemotherapy for other malignant diseases within the previous 5 years, except for neoadjuvant pre-cystectomy chemotherapy or adjuvant chemotherapy which are permitted.
8. Patients with the following severe acute co-morbidity are not eligible:

   * Unstable angina or congestive heart failure that required hospitalization in the 6 months before randomisation.
   * Transmural myocardial infarction in the 6 months prior to randomisation.
   * Acute bacterial or fungal infection requiring intravenous antibiotics at randomisation.
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of randomisation.
   * Severe hepatic disease: Child-Pugh Class B or C hepatic disease.
   * Known acquired immune deficiency syndrome (AIDS); the study treatment could impact blood count.
9. Patients with any other disease or illness which requires hospitalization or is incompatible with the study treatment are not eligible.
10. Patients unable to comply with study obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the study.
11. Patients enrolled in another therapeutic study within 30 days prior of randomisation.
12. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
pelvic recurrence-free survival (PRFS) | 3 years
  The PRFS is defined as the delay between randomization and pelvic recurrence or death, whichever occurs first. The pelvic recurrence will be evaluated according to RECIST V1.1 criteria.

SECONDARY OUTCOMES:
pelvic recurrence-free survival (PRFS) | 5 years
  The PRFS is defined as the delay between randomization and pelvic recurrence or death, whichever occurs first. The pelvic recurrence will be evaluated according to RECIST V1.1 criteria.
Disease-free survival (DFS) | 3 years
  DFS is defined as the delay between randomization and tumor progression (local, regional, or distant) or death of any cause, whichever occurs first.
Disease-free survival (DFS) | 5 years
  DFS is defined as the delay between randomization and tumor progression (local, regional, or distant) or death of any cause, whichever occurs first.
Overall Survival (OS) | 3 years
  OS is defined as the delay between randomization and death, of any cause.
Overall Survival (OS) | 5 years
  OS is defined as the delay between randomization and death, of any cause.
Metastasis-free survival (MFS) | 3 years
  MFS is defined as the delay between randomization, and metastasis (clinical or radiological) or death of any cause whichever occurs first.
Metastasis-free survival (MFS) | 5 years
  MFS is defined as the delay between randomization, and metastasis (clinical or radiological) or death of any cause whichever occurs first.
Disease-specific survival (DSS) | 3 years
  DSS is defined as the delay between randomization and death due to bladder cancer.
Disease-specific survival (DSS) | 5 years
  DSS is defined as the delay between randomization and death due to bladder cancer.
Tolerance will be evaluated by toxicity: acute (<6 months after RT) and late (≥6 months after RT), assessed using the NCI CTCAE Version N°4.0 | 5 years
  The tolerance will be evaluated by toxicity: acute (<6 months after RT) and late (≥6 months after RT), assessed using the NCI CTCAE Version N°4.0.
Patients' quality of Life | 5 years
  EORTC QLQ-C30
Patient quality of Life | 5 years
  The Bladder Cancer Index (BCI)
Evaluation of acute and late toxicities | 5 years
  The safety will be evaluated by toxicity: acute (<6 months after RT) and late (≥6 months after RT), assessed using the NCI CTCAE Version N°4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Paul SARGOS, MD, Principal Investigator — Institut Bergonié; Stéphane LARRE, Prof, Principal Investigator — CHU Robert Debré; Géraldine PIGNOT, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (17):
- France (17):
  - ICO Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Georges-Francois Leclerc, Dijon
  - Chu Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Hôpital Universitaire Dupuytren, Limoges
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - Saint Louis, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Chp Saint-Gregoire, Saint-Grégoire
  - ICO - site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse